CLINICAL TRIAL: NCT02784860
Title: Investigation of the Effects of Intravenous Lidocaine Infusion During Sedation for Colonoscopy
Brief Title: Effects of Intravenous Lidocaine During Sedation for Colonoscopy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor and Chair, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LIDOCOLO2016JJCF
Record Dates: First submitted 2016-05-02; First posted 2016-05-27 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Colonoscopy
Keywords: colonoscopy; lidocaine; propofol; sedation
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine. Administration of lidocaine is started with 1.5 mg/kg bolus injection followed by a continuous infusion of 4mg/kg/h.
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Placebo Administration of normal saline: same volume of saline as lidocaine.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Lidocaine — Propofol (0.5 mg/kg or more) is titrated to provide loss of consciousness. Then in the lidocaine group, lidocaine 2% is administered as a bolus followed by a continuous intravenous infusion after loss of consciousness
  Other Names: XYLOCAINE ; (NDA) 006488
  Arms: Lidocaine
Drug: normal saline — Propofol (0.5 mg/kg or more) is titrated to provide loss of consciousness. Then in the placebo group, the same volume of normal saline is administered after loss of consciousness
  Arms: Placebo

SUMMARY:
This study assesses the benefits of continuous intravenous lidocaine administration during sedation for colonoscopy.

Sedation will consist of propofol infusion titrated to provide adequate working conditions to the gastroenterologist. Patients will be randomly allocated into two groups: lidocaine infusion (bolus of 1.5 mg/kg followed by a continuous infusion of 4 mg/kg/h) or the same volume of placebo (normal saline)

DETAILED DESCRIPTION:
The potential benefits of lidocaine infusion will be tested on:

* propofol consumption (primary outcome)
* intraoperative respiratory depression
* time for patient recovery
* postoperative fatigue
* postoperative pain
* postoperative cognitive dysfunction

ELIGIBILITY:
Inclusion Criteria:

* colonoscopy without gastroscopy

Exclusion Criteria:

* lidocaine allergy
* epilepsy
* severe heart rhythm disorders
* renal failure with creatinine clearance lower than 30ml/minute

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Consumption of propofol | intraoperative
  Dose of propofol administered during sedation if measured at the end of it.

SECONDARY OUTCOMES:
Episodes of oxygen desaturation | intraoperative
  Episodes of oxygen desaturation: SpO2 < 95 and 90%
Time for recovery | intraoperative
  the patient is discharged when conscious and able to give his birth date
Quality of working conditions assessed by the gastroenterologist | intraoperative
Abdominal discomfort | intraoperative and 15 minutes later
  Evaluation with VAS (visual analog scale) form 0 (no discomfort) to 10 (unbearable Abdominal discomfort assessed on a 0 to 10 visual analog scale
Postoperative fatigue | 15 min after sedation
  Fatigue will be assessed on a visual analog scale
Cognitive condition | 15 minutes after sedation
  Cognitive condition will be evaluated with the MMSE (Minimal Mental State Examination)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Joris, MD, Principal Investigator — University of Liege
Locations (1):
- University Hospital of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forster C, Vanhaudenhuyse A, Gast P, Louis E, Hick G, Brichant JF, Joris J. Intravenous infusion of lidocaine significantly reduces propofol dose for colonoscopy: a randomised placebo-controlled study. Br J Anaesth. 2018 Nov;121(5):1059-1064. doi: 10.1016/j.bja.2018.06.019. Epub 2018 Aug 1. PMID 30336850